CLINICAL TRIAL: NCT03494478
Title: Emotional Dysregulation and Cyclothymia in Adult Patients With ADHD: Cohort Follow-up of Patients in Two Referral Centers
Brief Title: Emotional Dysregulation in Adult ADHD.
Acronym: EMO-TDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6795
Record Dates: First submitted 2018-03-23; First posted 2018-04-11 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Adult ADHD
Keywords: Cohort study; Emotion dysregulation; Questionnaires; Actimetry; Neuropsychology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort group (Experimental): All participants will have evaluations at inclusion and 12 months. Neuropsychological testing Actimetry Selfquestionnaires on emotional topics
  Interventions: Other: Neuropsychological testing; Other: Actimetry; Other: Self-questionnaires on emotional topics

INTERVENTIONS:
Other: Neuropsychological testing — The assessment will will be done at the time of the initial evaluation (undiagnosed / untreated patients), then at one year of follow-up
  Other Names: attention; working memory; executive functions
Other: Actimetry — The assessment will will be done at the time of the initial evaluation (undiagnosed / untreated patients), then at one year of follow-up.
  Other Names: Selfquestionnaires on emotional topics
Other: Self-questionnaires on emotional topics — The assessment will will be done at the time of the initial evaluation (undiagnosed / untreated patients), then at one year of follow-up.

SUMMARY:
Attention deficit disorder in adults with or without hyperactivity (ADHD) is a common disorder, affecting around 3% of the population. ADHD increases the risk of psychiatric disorders (mood disorders, sleep disorders, personality disorders, addictive behavior), risky behaviors, and vocational difficulties. Emotional dysregulation (ED) constitute a major hindrance in the daily life of subjects, with a great impact on the general functioning and the quality of life of the patients.

The investigators want to determine the characteristics of patients with each type of ED (impulsivity, exacerbated emotional intensity, cyclothymia, borderline personality traits), and study the stability of these traits over time. Since circadian rhythms influence mood and circadian rhythms frequently occur in patients with ADHD, the investigators want to determine if there is a link between ED and instability in circadian rhythms. Finally, they would like to observe whether the ED evolves and according to whether or not treatment is taken

ELIGIBILITY:
Inclusion criteria:

* Male or female aged ≥ 18 years
* diagnosis of adult ADHD prior to inclusion
* Affiliated to a social health insurance
* Subject having dated and signed informed consent
* Subject having been informed of the results of the prior medical examination

Exclusion criteria:

* Mobility project preventing follow-up for 1 year (planned move)
* impossibility to give the subject information enlightened (subject in emergency situation, difficulties in understanding the subject, mental retardation, illiteracy or insufficient command of the French language ...)
* Subject under the protection of justice
* Subject under guardianship or curatorship
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At inclusion
  Score of cyclothymia (TEMPS-A scale)
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At 12 months after inclusion
  Score of cyclothymia (TEMPS-A scale)
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At inclusion
  Score of emotional lability (ALS scale)
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At 12 months after inclusion
  Score of emotional lability (ALS scale)
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At inclusion
  Score of emotional dysregulation (WRAADDS scale)
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At 12 months after inclusion
  Score of emotional dysregulation (WRAADDS scale)
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At inclusion
  Score of borderline personality symptoms (BSL scale)
Characterization of emotional dysregulation (descriptive analysis of different scales assessing emotional dysregulation) | At 12 months after inclusion
  Score of borderline personality symptoms (BSL scale)

SECONDARY OUTCOMES:
Association between emotional dysregulation, cognitive deficits and circadian instability | At inclusion
  Correlation between emotional dysregulation and executive and attentional dysfunction measured with the TAP test.
  Correlation between emotional dysregulation and instability index of circadian rhythms measured by actimetry.
Association between emotional dysregulation, cognitive deficits and circadian instability | At 12 months after inclusion
  Correlation between emotional dysregulation and executive and attentional dysfunction measured with the TAP test.
  Correlation between emotional dysregulation and instability index of circadian rhythms measured by actimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien WEIBEL, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Centre Hospitalier Spécialisé de Rouffach - Secteur 8, Rouffach
  - Hôpitaux Universitaires de Strasbourg - Service de Psyhciatrie 2/PPSAM, Strasbourg

IPD SHARING:
Plan to Share IPD: No